CLINICAL TRIAL: NCT07015008
Title: Relationship Between Sleep Time and Maximal Fat Oxidation Capacity During Exercise.
Brief Title: Sleep and Maximal Fat Oxidation
Acronym: Sleep&Fat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Alberto Pérez-López, Principal Investigator, University of Alcala
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: CEID/2023/6/119_2
Record Dates: First submitted 2025-05-23; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Sleep Deprivation
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 8h Sleep (at home) (Placebo Comparator): Arm Description: Participants sleep 8h at home
  Interventions: Behavioral: Sleep deprivation; Behavioral: Sleep place
- 8h Sleep (Laboratory) (Experimental): Participants sleep 8h in the lab
  Interventions: Behavioral: Sleep deprivation; Behavioral: Sleep place
- 4h Sleep (Laboratory) (Experimental): Participants sleep 4h in the laboratory
  Interventions: Behavioral: Sleep deprivation
- 0h Sleep (Laboratory) (Experimental): Participants sleep 0h in the laboratory
  Interventions: Behavioral: Sleep deprivation

INTERVENTIONS:
Behavioral: Sleep deprivation — Partial (4h) or total (0h) sleep deprivation
Behavioral: Sleep place — 8h sleep at home or in the laboratory
  Arms: 8h Sleep (Laboratory); 8h Sleep (at home)

SUMMARY:
Introduction: Despite the awareness of the importance of sleep in our lives, especially for athletes, the consequences of poor rest on sports performance are not well understood. Furthermore, the interaction between complete and partial sleep deprivation over one night and sleeping the usual hours for each person remains unclear.

Objectives: The aim of this study is to evaluate the effects of sleep deprivation on maximal fat oxidation (MFO) in male and female participants.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:

  * Age between 18 and 35 years.
  * Body Mass Index (BMI) < 25 kg/m².
  * Resistance-trained individuals (more than 2 years of structured training).
  * Healthy men and women without neurological, cardiometabolic, immunological, or physical conditions that prevent them from exercising.
  * Participants must be able to perform the tests described in the following section.

Exclusion Criteria:

* History of neuromuscular diseases, heart disease, or conditions that may affect liver or muscle metabolism.
* Use of drugs, stimulants, or sports supplements that could interfere with the dietary supplement used in the study.
* Sedentary habits (less than 150 minutes/week of moderate exercise).
* Having undergone prolonged periods of physical inactivity in the 6 months prior to the study.
* Engaging in strenuous exercise within 48 hours prior to the tests.
* Failure to replicate the same food intake on both experimental days.
* Consumption of caffeine or any other stimulant the day before the tests.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Maximal Fat Oxidation Rate | Through study completion, an average of 4 weeks
  g/min using a metabolic chart

SECONDARY OUTCOMES:
Fat mass | Through study completion, an average of 4 weeks
  Using electrical bioimpedance (kg of body mass)
Fat-free mass | Through study completion, an average of 4 weeks
  Using electrical bioimpedance (kg of body mass)

CONTACTS AND LOCATIONS:
Locations (1):
- Facultad de Medicina y Ciencias de la Salud. Universidad de Alcalá, Alcalá de Henares, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes